CLINICAL TRIAL: NCT05920486
Title: The Effectiveness of High-Intensity Laser Therapy in Reducing Pain and Improving Function in Patients With Sacroiliitis: A Sham-Controlled Randomized Trial
Brief Title: High-Intensity Laser Therapy in Patients With Sacroiliitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 012/020230607
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Sacroiliac Arthritis
MeSH Terms: conditions — Arthritis, Sacroiliac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Laser Therapy (HILT) Group (Experimental): Participants in the HILT group will receive an 8-week course of High-Intensity Laser Therapy (HILT) for the treatment of sacroiliitis. HILT will be administered using a Class IV laser with a wavelength of 980 nm, power output of 10 W, spot size of 0.5 cm, and a dose of 60 J/cm2 per session. The laser will be applied to the affected area of the sacroiliac joint, with the aim of achieving a sensation of warmth in the region. The treatment sessions will be delivered for 10 minutes per session, with a total of 12 sessions over 8 weeks. Participants will receive no other specific interventions during the study period.
  Interventions: Device: High-Intensity Laser Therapy (HILT)
- Sham-Control Group (Sham Comparator): Participants in the sham-control group will receive a sham HILT treatment for the treatment of sacroiliitis. The sham treatment will be delivered using a device that looks like the HILT device, but does not emit laser energy. The device will be applied to the affected area of the sacroiliac joint, with the aim of achieving a sensation of warmth in the region. The treatment sessions will be delivered for 10 minutes per session, with a total of 12 sessions over 8 weeks. Participants will receive no other specific interventions during the study period.
  Interventions: Device: Sham High-Intensity Laser Therapy (HILT)

INTERVENTIONS:
Device: High-Intensity Laser Therapy (HILT) — High-Intensity Laser Therapy (HILT) is a non-invasive treatment that utilizes high-powered lasers to deliver therapeutic doses of energy to damaged tissue. In this study, HILT will be used to treat sacroiliitis, a condition that affects the sacroiliac joint in the lower back and pelvis. HILT will be administered using a Class IV laser with a wavelength of 980 nm, power output of 10 W, spot size of 0.5 cm, and a dose of 60 J/cm2 per session. The laser will be applied to the affected area of the sacroiliac joint, with the aim of achieving a sensation of warmth in the region. The treatment sessions will be delivered for 10 minutes per session, with a total of 12 sessions over 8 weeks. The aim of HILT is to promote cellular repair and regeneration, reduce pain, and improve function in patients with sacroiliitis. Participants in the HILT group will receive HILT treatment as the primary intervention in this study.
  Arms: High-Intensity Laser Therapy (HILT) Group
Device: Sham High-Intensity Laser Therapy (HILT) — Sham HILT is a non-invasive treatment that mimics the appearance and sensation of HILT but does not deliver any laser energy to the affected tissue. In this study, Sham HILT will be used as a control intervention for the treatment of sacroiliitis. The device used for Sham HILT will look and feel the same as the HILT device, but will not emit any laser energy. The device will be applied to the affected area of the sacroiliac joint, with the aim of achieving a sensation of warmth in the region. The treatment sessions will be delivered for 10 minutes per session, with a total of 12 sessions over 8 weeks. The aim of Sham HILT is to provide a credible control intervention that does not have any specific therapeutic effect on the sacroiliac joint. Participants in the Sham HILT group will receive Sham HILT treatment as the primary intervention in this study.
  Arms: Sham-Control Group

SUMMARY:
To investigate the effectiveness of High-Intensity Laser Therapy (HILT) in reducing pain and improving function in patients with sacroiliitis, aged 40-60 years.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults aged 40-60 years old
* Diagnosis: Confirmed diagnosis of sacroiliitis by a specialist (e.g., rheumatologist, orthopedic surgeon, or radiologist) based on a combination of clinical findings, laboratory tests, and imaging studies
* Clinical findings: Presence of at least one or more of the following clinical signs and symptoms suggestive of sacroiliitis:

  1. Low back pain, buttock pain, or hip pain, worsened by prolonged sitting, standing, or walking
  2. Stiffness in the lower back, buttock, or hip region, particularly in the morning or following prolonged inactivity
  3. Pain improvement with physical activity or exercise
* Duration of symptoms: Experiencing symptoms for at least 3 months

Exclusion Criteria:

* Previous surgery or invasive procedures targeting the sacroiliac joints
* Contraindications to physical interventions (e.g., spinal instability, fractures, or severe neurological deficits)
* Presence of other spinal pathologies or systemic inflammatory conditions that could confound the assessment of sacroiliitis (e.g., lumbar disc herniation, ankylosing spondylitis, or rheumatoid arthritis)
* Pregnant or breastfeeding women

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-06-22 (Estimated); Primary Completion 2024-03-22 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain intensity | Changes in Pain intensity Measured at baseline, week 4, week 8 (end of treatment), and week 12 (follow-up)
  The Numeric Pain Rating Scale is a self-reported measure of pain intensity, with a score ranging from 0 (no pain) to 10 (worst pain imaginable). Participants will be asked to rate their pain intensity at rest and during movement of the sacroiliac joint.
Changes in Functional ability | Changes in Functional ability Measured at baseline, week 4, week 8 (end of treatment), and week 12 (follow-up)
  The Oswestry Disability Index is a self-reported measure of functional ability, with a score ranging from 0% (no disability) to 100% (maximum disability). Participants will be asked to complete a questionnaire assessing their ability to perform various activities of daily living, such as walking, sitting, and standing.

SECONDARY OUTCOMES:
Global Perceived Effect (Global Perceived Effect Scale) | Measured at week 8 and week 12 (follow-up)
  The Global Perceived Effect Scale is a self-reported measure of the participant's overall improvement, with a score ranging from -5 (vastly worse) to 5 (completely recovered). Participants will be asked to rate their perceived overall improvement in their condition.
Changes in Range of Motion in the Lumbopelvic Region (Modified Schober Test and Hip Flexion/Extension) | Changes in Range of Motion Measured at baseline, week 4, week 8 (end of treatment), and week 12 (follow-up)
  The Modified Schober Test is an objective measure of lumbar flexion, and the Hip Flexion/Extension Test is an objective measure of hip range of motion. These tests will be used to assess changes in range of motion in the lumbopelvic region following the intervention.
Changes in Health-Related Quality of Life (Short Form 36 Health Survey) | Changes in Health-Related Quality of Life Measured at baseline, week 4, week 8 (end of treatment), and week 12 (follow-up)
  The Short Form 36 Health Survey is a self-reported measure of health-related quality of life, consisting of 36 items that assess various aspects of physical and mental health. The survey yields scores on eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Cairo University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No